| The Effectiveness of the Video Conferencing Telerehabilitation Method, Delivered in One on One and Group Sessions, in Urinary Incontinence Cases. |
|---|
| Study Protocol and Statistical Analysis Plan (SAP) (Pages 1 – 21) |
| November 15,2021 |

#### The Effectiveness of the Video Conferencing

# Telerehabilitation Method, Delivered in One on One and Group Sessions, in Urinary Incontinence Cases.

**Study Protocol (Pages 2-6)** 

**November 15,2021** 

#### **Study Protocol**

Study titled "The Effectiveness of the Video Conferencing Telerehabilitation Method, Delivered in One on One and Group Sessions, in Urinary Incontinence Cases." was approved by Marmara University Faculty of Medicine Ethical Committee at the meeting on 30.11.2020 with approval number: 1195 (Annex-1).

The legal representatives of the patients who participated in the study will be informed about the aim, duration and the programs to be applied throughout the study. Volunteer Information Form will be signed and approved in accordance with the standards deemed appropriate by the Ethical Committee of Marmara University Faculty of Medicine. The study will be conducted in accordance with the Declaration of Helsinki.

#### **Hypothesis of the Study**

**H0:** With one on one video conference method, exercise training is no superiority of exercise training with group video conferencing method in urinary incontinence.

**H1:** Exercise training with one on one video conference method is more effective in increasing muscle strength in patients with urinary incontinence.

**H2**: One on one videoconferencing and exercise training are more effective in reducing the degree of incontinence in patients with urinary incontinence.

**H3:** Exercise training with one on one videoconferencing method is more effective in increasing the quality of life in patients with urinary incontinence.

**H4:** Exercise training with one on one videoconferencing method is more effective in increasing patient satisfaction in patients with urinary incontinence.

**H5:** Exercise training with one on one video conference method is more effective in increasing sexual function in patients with urinary incontinence.

**H6:** Exercise training with one on one videoconferencing method is more effective in increasing exercise adherence in patients with urinary incontinence.

#### Randomization of the Study Groups

Individuals with Urinary İncontinence applying to Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi will be invited to participate in the study. Individuals who volunteered to participate and whom met the criteria for participation will be randomized with simple random sampling method and will be

divided into two groups. In both groups participants will receive same exercise program and physiotherapist will follow up the exercise program every week by video confernce method. While only the physiotherapist and the patient will take part in the one-on-one group, there will be a physiotherapist and 8 patients in the group sessions.

#### **Inclusion Criteria**

18-65 aged

BMI 18-30 kg/m2

Being diagnosed with stress incontinence or mixed incontinence (dominantly SUI)

Mild or moderate incontinence (mild SUI; urinary incontinence with coughing, sneezing, laughing, or any strenuous activity. Moderate; urinary incontinence with carrying, pushing, lifting, walking, and any light physical activity)

#### **Exclusion Criteria**

Pregnancy

Ongoing vulvovaginitis or urinary tract infection or malignancy

Pelvic floor muscle strength is between 0-1 according to the Modified Oxford Scale,

Previous surgery for SUI

Problems with vision or inability to understand given commands

Conservative therapy in the last 6 months

Allergic reaction to the gel used with the perinometer/probe

#### **Evaluations**

Evaluation parameters will be applied at the baseline, at the end of 4-weeks treatment program, at the end of 8 weeks treatment program. Outcome measures and applied evaluations are shown in Table 1.

**Table 1.** Outcome measures and evaluation methods

| Primary Outcome<br>Measures | Evaluation Methods |
|-----------------------------|---------------------------|
| | -PERFECT Scheme |
| Muscle Strength | -Surface Electromyography |

| Secondary Outcome | Evaluation Methods |
|---|---|
| Measures | Evaluation Methods |
| | -1 hour pad test |
| | -The International Consultation on Incontinence Questionnaire-<br>Short Form |
| Symptom Evaluation | - Urogenital Distress Inventory- 6 (UDI-6) |
| | - Incontinence Impact Questionnaire-7 (IIQ-7) |
| | - Overactive Bladder -Validated 8- Question Awereness Tool (OAB-V8) |
| Patient Satisfaction | Visual Analog Scale (VAS) |
| Exercise Adherence | VAS Broome Pelvic Floor Muscle Exercise Self- Efficiacy Scale |
| Sexual Function | Female Sexual Function Scale (FSFI) |

#### **Treatment Program**

The exercises which given the both groups compose same exercise protocols for 8 week. The exercise protocol includes pelvic floor muscle training, diaphragmatic breathing exercise and core exercise will be given the all participants. The participants in the study will be followed up with video conferecing method by weekly.

**Group I (one on one video conferencing group):** In this group, exercise follow-up and transition to the next exercise phase will be realized with one-on-one video conference interviews.

**Group II (group sessions video conferencing group):** In this group, exercise follow-up and transition to the next exercise stage will be realized with group video conference sessions consisting of 8 participants.

| The Effectiveness of the Video Conferencing Telerehabilitation Method, Delivered in One on One and Group Sessions, in Urinary Incontinence Cases. |
|---|
| Statistical Analysis Plan (SAP) (Pages 7 –8) |
| November 15,2021 |

#### **Statatistical Analysis Plan (SAP)**

In the analysis of the data to be obtained in the study, the significance will be evaluated at the p<0.05 level with the SPSS 22.0 statistical program at the 90% confidence interval. In the evaluation of variables; If the number of cases is sufficient, its conformity to the normal distribution will be questioned with the Kolmogorov Smirnov test and normal distribution graphs. In the examination of the variables, appropriate statistical tests will be applied depending on the provision of parametric or non-parametric test conditions. Normally distributed variables will be expressed as mean and standard deviation, and non-normally distributed variables will be expressed as numbers and percentages. If the groups fit the normal distribution, the evaluation results at the beginning, 4th week and 8th week will be compared with ANOVA, if the normal distribution is not met, comparisons will be made with Kruskal Wallis and appropriate post-hoc tests. In the correlation analysis, the appropriate Speerman or Pearson correlation analysis methods will be preferred. Chi-square test will be used in the evaluation of binary data.

| The Effectiveness of the Video Conferencing Telerehabilitation Method, Delivered in One on |
|---|
| One and Group Sessions, in Urinary Incontinence Cases. |
| Annex (Pages 9 – 21) |

**November 15,2021** 

**Annex 1.** Marmara University Faculty of Medicine Ethical Committee Approval (Approval made at the meeting on 30.11.2020 with number: 1195)

| | | Marmara On<br>Klinik Araştı | iversites<br>rmalar I | i Tip Fi<br>Etik Ku | akültesi<br>rulu | | | |
|---|---|---|---|---|---|---|---|---|
| | PROTOKOL KODU | | | 21.119 | 5 | | | |
| | PROJE ADI SORUMLU ARAȘTIRICI ÜNVANI/ADI | | ÜRINER INKONTİNANSLI ÖLGULARDA BİRE BİR V<br>GRUP ŞEKLİNDE VERİLEN VİDEO KONFERAN<br>TELEREHABİLİTASYON YÖNTEMİNİN ETKİNLİĞİ<br>Doç. Dr. Aysel YILDIZ ÖZER | | | | | |
| CARAR BILGILERI | maran increaming to gerrak! | eştirilmesinde sakıncı<br>i proje değişiklikleri | a butonmad | fulls icim b | Corollomuses | E OMESSA | COLUMN DESCRIPTION OF THE PERSON OF THE PERS | sç, yaklaşım ve yüstemleri dikk<br>diriği ile karac verilmiştir. O<br>nin Etik Karula bildirilerek pi |
| TELER<br>Unvani / Adi / Seyadi | Uzmanlık Dalı | Kurumu / EK Üyel | ligi | | inan Proje<br>Hiskisi | | fantiya<br>itdus | Imea |
| Prof.Dr. Haner DİRESKENELİ | Ramateleji | M.Ü Tıp Fakültes | i/Başkan | Var | Yok | Evet | Hayır | 1 |
| Prof.Dr. Tillin ERGUN | Dermatoloji | M.Ö Tıp Fakültes<br>Yrd. | si/Başkan | Var | Yok | Evet | Hayır | \$ |
| Prof.Dr. Asile KARAALP | Farmakoloji | M.O Tip Fakült | tesi/Oye | Var | Yok | EVET | HAYIR | 1/, |
| Prof. Dr. Şelik GÖRKEY | Tip Tarihi ve Etik | MLC Top Faktin | test/Oye | Var | Yok | Evet | Hayir | 1 from |
| Prof.Dr. Handan KAYA | Patoloji | M.O Top Fakült | tesi/Oye | Var | Yok | Evet | Hayır | 1000 |
| Prof.Dr. M.Bahader GÜLLÜÖĞL | .U Genel Cerrahi | M.O Top Faktio | tesi/Üye | Var | Yok | Evet | Hayır | My |
| Prof.Dr. Semra SARDAŞ | Еслис | M.Ü Eczacilik F | ak/Üye | Var | Yok | Evet | Hayır | 100 |
| Prof.Dr. Bajak DOĞAN | Dip Hekimi | M.Ü Diş Hekimliğ | i Fak/Üye | Var | Yok | Evet | Hayır | 1/95 |
| Prof. Dr. Beste Melek ATASOY | Radyusyon<br>Onkolojisi | M.O Top Fakille | tesi/Üye | Var | Yok | Evet | Hayır | X |
| Prof. Dr., EBF KARAKOÇ<br>AYDINER | Çocuk Sağlığı ve<br>Hastalıkları | M.O Tip Faküli | tesi/Üye | Var | Yok | Evet | Hayır | The same |
| ProfDr. Meltem KORAY | Dis Hekimi | İstanbul Üniv. Diş<br>Fak/Üye | | Var | Yok | Evet | Hayır | |
| Doç. Dr. Gürkan SERT | Hukukçu | 100000000000000000000000000000000000000 | | Var | Yok | Evet | Hayır | Br |
| Dog.Dr: Figra DEMİR | Halk Sağlığı | Acıbadem Üniv. | Tip Fak. | Var | Yok | Evet | Hayır | |
| Dog.Dr. Pinar Mega TİBER | Biyoficik | M.O Tip Faksii | tesi/Oye | Var | Yok | Evet | Hayır | U. |
| Glade Ayour MİRZA | Sağlık Mensubu<br>olmayan kişi | Serbest | | Var Y | ok O | Evet | Hayır | |

#### **Annex 2. Patient Evaluation Form**

| PATİENT | EVALUATION | FORM | DATE: |
|------------------------------|------------|---------------|-------|
| NAME-SURNAME: | | | |
| SEX: | | | |
| BİRTH DATE/AGE: | | | |
| HEIGHT: | WEIGHT: | | BMI: |
| EDUCATION LEVEL: | | | |
| MARITUAL STATUS: | | | |
| PHONE NUMBER: | | | |
| NUMBER OF BİRTH: | | TYPE OF BİRTH | : |
| MENOPEASE STATUS: | | | |
| WEEKLY ALCOHOL CONSUMPTION: | / week | | |
| WEEKLY TEA CONSUMPTION: | | | |
| WEEKLY CAFFEINE CONSUMPTION: | / week | | |
| MEDİCAL HİSTORY: | | | |
| DRUGS USED: | | | |

### Annex 3. Assessment of Muscle Strength

| | PERFECT SCHEME | | | | |
|---|---|---|---|---|---|
| | Power | Endurance | Repetitions | Fast Contraction | Every Contraction Time |
| | (P) | (E) | (R) | (F) | (ECT) |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| MEAN | | | | | |

| Surface EMG | | | |
|-------------|---------|-------------|------------------|
| | | Maximum | |
| | Resting | Voluntary | Pelvic Floor |
| | tone | Contraction | Muscle Endurance |
| | | (MVC) | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| Mean | | | |

# Annex 4. International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form

| | | ICIQ-UI Short Form | |
|---|---|---|---|
| Initi | ial number | CONFIDENTIAL | DAY MONTH<br><b>Today's da</b> |
| and | d how much this bothers | them. We would be grat | to find out how many people lead<br>eful if you could answer the fo<br>ge, over the PAST FOUR WEEKS |
| 1 | Please write in your date | of birth: | DAY MONTH YE |
| 2 | Are you (tick one): | | Female Male |
| 3 | How often do you leak uri | ine? (Tick one box) | |
| | | | never |
| | | abo | ut once a week or less often |
| | | | two or three times a week |
| | | | about once a day several times a day |
| | | | all the time |
| - | We would like to know ho<br>How much urine do you <u>u</u><br>(Tick one box) | | leaks. |
| - | How much urine do you <u>u</u> | | leaks. wear protection or not)? |
| 5 ( | How much urine do you <u>u</u> | usually leak (whether you | leaks. none none a small amount a moderate amount a large amount th your everyday life? |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between | usually leak (whether you | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between | leaking urine interfere wieen 0 (not at all) and 10 (a | leaks. none none a small amount a moderate amount a large amount th your everyday life? great deal) 7 8 9 10 |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between | leaking urine interfere wi<br>een 0 (not at all) and 10 (a<br>2 3 4 5 6 7 | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 7 8 9 10 a great deal score: sum scores 3+4+5 |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between the second sec | leaking urine interfere wieen 0 (not at all) and 10 (a 2 3 4 5 6 7 ICIQ | leaks. I wear protection or not)? none a small amount a moderate amount a large amount th your everyday life? great deal) 7 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between the second sec | leaking urine interfere wileen 0 (not at all) and 10 (a 2 3 4 5 6 7 ICIQ | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak fore you can get to the toilet |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between the second sec | leaking urine interfere wileen 0 (not at all) and 10 (a 2 3 4 5 6 7 ICIQ | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 7 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak fore you can get to the toilet s when you cough or sneeze |
| 5 ( | How much urine do you u (Tick one box) Overall, how much does I Please ring a number between the second sec | leaking urine interfere wileen 0 (not at all) and 10 (a 2 3 4 5 6 7 ICIQ Please tick all that apply to leaks be leaks | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak fore you can get to the toilet |
| 5 ( | How much urine do you under (Tick one box) Overall, how much does It Please ring a number between the properties of the | leaking urine interfere will een 0 (not at all) and 10 (a 2 3 4 5 6 To lCIQ Please tick all that apply to leaks be leaks | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak fore you can get to the toilet s when you cough or sneeze leaks when you are asleep |
| 5 ( | How much urine do you under (Tick one box) Overall, how much does It Please ring a number between the properties of the | leaking urine interfere will een 0 (not at all) and 10 (a 2 3 4 5 6 To lCIQ Please tick all that apply to leaks be leaks | leaks. none a small amount a moderate amount a large amount th your everyday life? great deal) 8 9 10 a great deal score: sum scores 3+4+5 you) never – urine does not leak fore you can get to the toilet swhen you cough or sneeze leaks when you are asleep e physically active/exercising |

Thank you very much for answering these questions.

Copyright © "ICIQ Group"

#### Annex 5. Urogenital Distress Inventory (Udi 6)

### **UROGENITAL DISTRESS INVENTORY (UDI 6)**

Do you experience? If so how much are you bothered by:

| | Not at all | A little bit | Moderately | Greatly |
|---|---|---|---|---|
| 1. Frequent urination? | 0 | 1 | 2 | 3 |
| 2. Urine leakage related to the feeling of urgency? | 0 | 1 | 2 | 3 |
| 3. Urine leakage related to physical activity, coughing or sneezing? | 0 | 1 | 2 | 3 |
| 4. Small amounts of urine leakage (that is drops)? | 0 | 1 | 2 | 3 |
| 5. Difficulty emptying your bladder? | 0 | 1 | 2 | 3 |
| 6. Pain or discomfort in the lower abdominal or genital area? | 0 | 1 | 2 | 3 |

#### Annex 6. Incontinence Impact Questionnaire, Short Form (Iiq-7)

| OREGON HEALTH OF SUIT | Patient Name: Date of Birth: MRN: Date of Service: Physician: |
|---|---|
|---|---|

#### **Incontinence Impact Questionnaire, Short Form (IIQ-7)**

Some people find that accidental urine loss may affect their activities, relationships, and feelings. For each question, circle the response that best describes how much your activities, relationships, and feelings are being affected by urine leakage over the past month.

#### Has urine leakage (incontinence) affected your:

| | Not at All | Slightly | Moderately | Greatly |
|---|---|---|---|---|
| Ability to do household chores (cooking, housecleaning, laundry)? | 0 | 1 | 2 | 3 |
| Physical recreation such as walking, swimming, or other exercise? | 0 | 1 | 2 | 3 |
| Entertaining activities (movies, concerts, etc.)? | 0 | 1 | 2 | 3 |
| Ability to travel by car or bus more than 30 minutes from home? | 0 | 1 | 2 | 3 |
| Participation in social activities outside your home? | 0 | 1 | 2 | 3 |
| Emotional health (nervousness, depression, etc.)? | 0 | 1 | 2 | 3 |
| Feeling frustrated? | | | | |
| | 0 | 1 | 2 | 3 |

Adapted from Uebersax JS, Wyman FF, Shumaker SA, et al. Short forms to assess life quality and symptom distress for urinary incontinence in women: the incontinence impact questionnaire and urogenital distress inventory. Neurourol Urodyn 1995; 14: 131.

#### **Annex 7. Assessment of Patient Satisfaction**

| 1) How satisfied were yo | with the treatment you rece | ived? |
|---|---|---|
| 0 | 5 | 10 |
| (Not satisfied at a | 11) | (Very satisfied) |
| 2) How satisfied were yo | a with the decrease in your co | omplaints after your treatment? |
| 0 | 5 | 10 |
| (Not satisfied at a | 11) | (Very satisfied) |
| 3) How satisfied were yo | ı that your exercise program | is followed by online interviews? |
| 0 | 5 | 10 |
| (Not satisfied at a | 11) | (Very satisfied) |

#### **Annex 8. Assesment of Exercise Adherence**

#### - Visual Analog Scale

| How long did you adher | e to the exercise program durin | g your treatment? |
|------------------------|---------------------------------|-------------------|
| 0 | 5 | 10 |
| (Not satisfied at | all) | (Very satisfied) |

#### - Broome Pelvic Muscle Exercise Self Efficiacy Scale

Level of Confidence Part A: How confident are you that you can: 1. Contract your pelvic muscles? 0 10 20 30 40 50 60 70 80 90 100 2. Perform pelvic muscle contractions three times a day? 0 10 20 30 40 50 60 70 80 90 100 3. Perform pelvic muscle contractions while lying down? 0 10 20 30 40 50 60 70 80 90 100 4. Perform pelvic muscle contractions while standing? 5. Perform pelvic muscle contractions while sitting? 0 10 20 30 40 50 60 70 80 90 100 0 10 20 30 40 50 60 70 80 90 100 6. Contract your pelvic muscles without contracting your abdominal muscles? 7. Contract your pelvic muscles while washing fruits under running water? 0 10 20 30 40 50 60 70 80 90 100 8. Contract your pelvic muscles when lifting a bag of groceries? 0 10 20 30 40 50 60 70 80 90 100 9. Contract your pelvic muscles while standing at the sink brushing your teeth? 0 10 20 30 40 50 60 70 80 90 100 0 10 20 30 40 50 60 70 80 90 100 10. Contract your pelvic muscles rapidly? 11. Perform pelvic muscle contractions when you are sad? 0 10 20 30 40 50 60 70 80 90 100 12. Contract your pelvic muscles while showering after a busy and tiring day? 0 10 20 30 40 50 60 70 80 90 100 13. Perform pelvic muscle contractions when you are tired? 0 10 20 30 40 50 60 70 80 90 100 14. Contract your pelvic muscles when you awaken at night with a strong urge to urinate? 0 10 20 30 40 50 60 70 80 90 100 Part B: How confident are you that pelvic muscle contractions will prevent unwanted urine loss: 1. When you experience a strong urge to urinate? 0 10 20 30 40 50 60 70 80 90 100 2. When you sneeze? 0 10 20 30 40 50 60 70 80 90 100 3. When you laugh? 0 10 20 30 40 50 60 70 80 90 100 4. While waiting 2 minutes for a restroom? 0 10 20 30 40 50 60 70 80 90 100 5. While waiting 5 minutes for a restroom? 0 10 20 30 40 50 60 70 80 90 100 6. When you wake up at night with a strong urge to urinate? 0 10 20 30 40 50 60 70 80 90 100 7. When you lift a heavy package? 0 10 20 30 40 50 60 70 80 90 100 0 10 20 30 40 50 60 70 80 90 100 8. When you cough? 9. When washing fruits and vegetables? 0 10 20 30 40 50 60 70 80 90 100

<sup>&</sup>lt;sup>a</sup> Reprinted, with permission of the publisher, the Society of Urologic Nurses and Associates Inc, from: Broome B. Psychometric analysis of the Broome Pelvic Muscle Self-Efficacy Scale in African-American women with incontinence. *Ural Nurs*. 2001;21:289–297.

#### **Annex 9. Female Sexual Function Index Score**

#### Question

Q1: Over the past 4 weeks, how often did you feel sexual desire or interest?

#### Response Options

5 = Almost always or always

4 = Most times (more than half the time)

3 = Sometimes (about half the time)

2 = A few times (less than half the time)

1 = Almost never or never

Q2: Over the past 4 weeks, how would you rate your **level** (degree) of sexual desire or interest?

5 = Very high

4 = High

3 = Moderate

2 = Low

1 = Very low or none at all

Q3. Over the past 4 weeks, how often did you feel sexually aroused ("turned on") during sexual activity or intercourse? 0 = No sexual activity

5 = Almost always or always

4 = Most times (more than half the time)

3 = Sometimes (about half the time)

2 = A few times (less than half the time)

1 = Almost never or never

Q4. Over the past 4 weeks, how would you rate your **level** of sexual arousal ("turn on") during sexual activity or intercourse?

0 = No sexual activity

5 = Very high

4 = High

3 = Moderate

2 = Low

1 = Very low or none at all

Q5. Over the past 4 weeks, how **confident** were you about becoming sexually aroused during sexual activity or intercourse?

0 = No sexual activity

5 = Very high confidence

4 = High confidence

3 = Moderate confidence

2 = Low confidence

1 = Very low or no confidence

Q6. Over the past 4 weeks, how **often** have you been satisfied with your arousal (excitement) during sexual activity or intercourse? Response Options 0 = No sexual activity

5 = Almost always or always

4 = Most times (more than half the time)

3 = Sometimes (about half the time)

2 = A few times (less than half the time)

1 = Almost never or never

- Q7: Over the past 4 weeks, how often did you become lubricated ("wet") during sexual activity or intercourse?
- 0 = No sexual activity
- 5 = Almost always or always
- 4 = Most times (more than half the time)
- 3 = Sometimes (about half the time)
- 2 = A few times (less than half the time)
- 1 = Almost never or never
- Q8. Over the past 4 weeks, how difficult was it to become lubricated ("wet") during sexual activity or intercourse?
- 0 = No sexual activity
- 1 = Extremely difficult or impossible
- 2 = Very difficult
- 3 = Difficult
- 4 = Slightly difficult
- 5 = Not difficult
- Q9: Over the past 4 weeks, how often did you main tain your lubrication ("wetness") until completion of sexual activity or intercourse?
- 0 = No sexual activity
- 5 = Almost always or always
- 4 = Most times (more than half the time)
- 3 = Sometimes (about half the time)
- 2 = A few times (less than half the time)
- 1 = Almost never or never
- Q10: Over the past 4 weeks, how **difficult** was it to maintain your lubrication ("wetness") until completion of sexual activity or intercourse?
- 0 = No sexual activity
- 1 = Extremely difficult or impossible
- 2 = Very difficult
- 3 = Difficult
- 4 = Slightly difficult
- 5 = Not difficult
- Q11. Over the past 4 weeks, when you had sexual stimulation or intercourse, how often did you reach orgasm (climax)?
- 0 = No sexual activity
- 5 = Almost always or always
- 4 = Most times (more than half the time)
- 3 = Sometimes (about half the time)
- 2 = A few times (less than half the time)
- 1 = Almost never or never
- Q12: Over the past 4 weeks, when you had sexual stimulation or intercourse, how **diffi**cult was it for you to reach orgasm (climax)?
- 0 = No sexual activity
- 1 = Extremely difficult or impossible
- 2 = Very difficult
- 3 = Difficult.
- 4 = Slightly difficult
- 5 = Not difficult
- Q13: Over the past 4 weeks, how satisfied were you with your ability to reach orgasm (climax) during sexual activity or intercourse?
- 0 = No sexual activity
- 5 = Very satisfied 4
- 4 = Moderately satisfied
- 3 = About equally satisfied and dissatisfied
- 2 = Moderately dissatisfied
- 1 = Very dissatisfied
- Q14: Over the past 4 weeks, how satisfied have you been with the amount of emotional closeness during sexual activity between you and your partner?
- 0 = No sexual activity
- 5 = Very satisfied
- 4 = Moderately satisfied
- 3 = About equally satisfied and dissatisfied
- 2 = Moderately dissatisfied
- 1 = Very dissatisfied

- Q15: Over the past 4 weeks, how satisfied have you been with your sexual relationship with your partner?
- 5 = Very satisfied
- 4 = Moderately satisfied
- 3 = About equally satisfied and dissatisfied
- 2 = Moderately dissatisfied
- 1 = Very dissatisfied
- Q16: Over the past 4 weeks, how satisfied have you been with your overall sexual life?
- 5 = Very satisfied
- 4 = Moderately satisfied
- 3 = About equally satisfied and dissatisfied
- 2 = Moderately dissatisfied
- 1 = Very dissatisfied
- Q17: Over the past 4 weeks, how often did you experience discomfort or pain during vaginal penetration?
- 0 = Did not attempt intercourse
- I = Almost always or always
- 2 = Most times (more than half the time)
- 3 = Sometimes (about half the time)
- 4 = A few times (less than half the time)
- 5 = Almost never or never
- Q18: Over the past 4 weeks, how often did you experience discomfort or pain following vaginal penetration?
- 0 = Did not attempt intercourse
- 1 = Almost always or always
- 2 = Most times (more than half the time)
- 3 = Sometimes (about half the time)
- 4 = A few times (less than half the time)
- 5 = Almost never or never
- Q19. Over the past 4 weeks, how would you rate your **level** (degree) of discomfort or pain during or following vaginal penetration?
- 0 = Did not attempt intercourse
- 1 = Very high
- 2 = High
- 3 = Moderate
- 4 = Low
- 5 = Very low or none at all

<sup>\*</sup> For the complete FSFI questionnaire, instructions and scoring algorithm, please see www.FSFkquestionnaire.com, or contact Raymond Rosen Ph.D., (Department of Psychiatry: UMDNJ-Robest Wood Johnson Medical School, 675 Hoes Lane, Piscataway, NJ 08854)

#### Annex 10. Overactive Bladder 8- Question Awereness Tool

# 0AB-**V**8

## Overactive Bladder-Validated 8-question Screener<sup>1</sup>

The questions below ask about how bothered you may be by some bladder symptoms. Some people are bothered by bladder symptoms and may not realize that there are treatments available for their symptoms. Please circle the number that best describes how much you have been bothered by each symptom. Add the numbers together for a total score and record the score in the box provided at the bottom.

| How bothered have you been by | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | A great<br>deal | A very<br>great deal |
|---|---|---|---|---|---|---|
| <ol> <li>Frequent urination during the daytime hours?</li> </ol> | 0 | 1 | 2 | 3 | 4 | 5 |
| 2. An uncomfortable urge to urinate? | 0 | 1 | 2 | 3 | 4 | 5 |
| 3. A sudden urge to urinate with little or no warning? | 0 | 1 | 2 | 3 | 4 | 5 |
| 4. Accidental loss of small amounts of urine? | 0 | 1 | 2 | 3 | 4 | 5 |
| 5. Nighttime urination? | 0 | 1 | 2 | 3 | 4 | 5 |
| 6. Waking up at night because you had to urinate? | 0 | 1 | 2 | 3 | 4 | 5 |
| 7. An uncontrollable urge to urinate? | 0 | 1 | 2 | 3 | 4 | 5 |
| 8. Urine loss associated with a strong desire to urinate? | 0 | 1 | 2 | 3 | 4 | 5 |
| Are you male? | If m | nale 🔲 a | dd 2 poi | nts to y | our score | <u> </u> |

| Please add up your responses to the questions above $lacksquare$ |
|------------------------------------------------------------------|
|------------------------------------------------------------------|

Please hand this page to your doctor when you see him/her for your visit.

If your score is 8 or greater, you may have overactive bladder. There are effective treatments for this condition. You may want to talk with a healthcare professional about your symptoms.

Note: You may be asked to give a urine sample. Please ask before going to the bathroom. Reference: 1. Data on file. Pfizer Inc, New York, NY.